CLINICAL TRIAL: NCT03135366
Title: Delivering Community-based Interventions and Disease Management Tools Across a Digital Platform in Order to Increase TB Treatment Adherence in LMICs
Brief Title: Self-verification and Support Via Mobile Phones Drastically Improves Tuberculosis Treatment Success in LMIC Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Keheala (Unknown); MIT's Applied Cooperation Team (Unknown); Kenya National Tuberculosis, Leprosy and Lung Disease Program (Unknown)
Responsible Party: Principal Investigator, Erez Yoeli, Research Scientist and Co-Director of the Applied Cooperation Team, Massachusetts Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HarvardU
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB; Adherence; Mobile Health; mHealth; Behavior change; Social and Behavior Change Communication (SBCC); Drug-Resistance; Keheala
MeSH Terms: conditions — Tuberculosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: We will employ a randomized controlled trial (RCT) with 600 patients included in the treatment group and 600 patients included in the control group. We have selected this methodology for the following reasons:
  1. RCTs are the gold-standard for providing evidence-based evaluation of medical interventions, and recommended when feasible.
  2. Keheala is a new program, and cannot be studied using existing data.
  3. We are working with researchers from Harvard's Program for Evolutionary Dynamics and Yale's Human Cooperation Lab, who have an established record of designing large-scale RCTs in real-world settings such as ours.
  This sample size was chosen to achieve 80% power in detecting improvements of 7.5% or more in the relevant health outcomes. To do this calculation, we employed Monte Carlo simulations of patient outcomes, based on the Kenyan Ministry of Health's 2013 TB Case Findings Report.
  Note: The sample size and outcomes were registered in December 2015 with the IRB.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Control) (Active Comparator)
  Interventions: Other: Standard of Care
- Keheala Intervention (Treatment) (Experimental): The intervention consisted of a daily request for self-verification of medication adherence, access to a supporter via a chat client, and information about TB.
  Interventions: Behavioral: Keheala

INTERVENTIONS:
Behavioral: Keheala
  Arms: Keheala Intervention (Treatment)
Other: Standard of Care — Patients receive medication for a week or two weeks at a time. They are assigned a friend or family member 'supporter' to verify the patient's at-home treatment and instructed to return to the clinic with the patient during medication refills.
  Arms: Standard of Care (Control)

SUMMARY:
Each year, 10.4 million patients are diagnosed with and 1.8 million people die from Tuberculosis (TB). Despite the availability of highly effective and accessible medications in the developing world where TB is endemic, the 6-18 month treatment regimen is often thwarted as patients fail to comply due to a lack of knowledge about the disease, desire for privacy, and/or stigma avoidance. Inappropriate medication use leading to multi-drug resistant (MDR) TB infects 5% of all TB patients, yet accounts for a significant proportion of all spending. In Kenya, the burden of TB is among the highest in the world with a prevalence rate of 558 cases per 100,000 people. There is a great need for the development of alternative protocols, which reduce the costs of treatment and burden of adherence, and more effectively motivate patients to adhere to the program. A substantial and growing literature in the social sciences demonstrates the potential of behavioral interventions for generating large increases in contributions to public goods.

This 1200 participant, Randomized Controlled Trial (RCT) explores the capacity of Keheala, a feature-phone and Internet-based digital platform that uses Unstructured Supplementary Service Data (USSD) technology, to deliver behavioral interventions for improving treatment adherence, outcomes and quality of life for TB patients in Nairobi, Kenya. Keheala taps into this underutilized potential by developing a powerful, cost-effective platform for better engaging patients' sense of responsibility to their community in order to increase adherence.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the deadliest infectious disease in the world. The latest estimates suggest there were 10.4 million cases in 2015 and 1.8 million TB deaths. Despite the availability of highly effective medications for treating TB in the developing world, lack of adherence to the treatment regimen remains the driving influence leading to multi-drug resistant (MDR) TB, morbidity and mortality. Conventional treatment is a lengthy process which depends heavily on patient adherence in seeking and then carrying out the prescribed treatment. Recognizing this challenge, the World Health Organization has developed a protocol for treating TB called Direct Observation of Treatments, Short-course (DOTS), but it is expensive and difficult to institute on a large-scale in resource-constrained regions, evidenced by its use in only 30% of all cases. This protocol also further burdens TB patients who are already some of the most marginalized individuals in society by requiring them to take time off from work in order to travel to the TB clinic for treatment verification. The patient may find this embarrassing if there is a stigma surrounding the disease in the community, or at the least, an unwelcomed intrusion into one's privacy. There is therefore great need for the development of alternative protocols, which reduce the costs of treatment and burden of adherence, and more effectively motivate patients to adhere to the program.

TB is spread through the air when people who are sick with TB excrete the causative bacillus, Mycobacterium tuberculosis mainly through coughing. Left untreated, a single patient can infect between 12 and 15 persons per year, a stark contrast to an Ebola patient who will only infect between 1.5 and 2.5 persons. When a patient adheres to the treatment regime, she makes it less likely that others will become sick, contributing to the health of her family and community. Adherence is thus a contribution to a public good--a personally costly action that benefits others. A substantial and growing literature in the social sciences demonstrates the potential of behavioral interventions for generating large increases in contributions to public goods, yet this potential has largely been left untapped in the treatment of TB. Keheala taps into this underutilized potential by developing a powerful, cost-effective platform for better engaging patients' sense of responsibility to their community in order to increase adherence.

Keheala is a feature-phone and Internet-based digital platform that uses text message-like interactions to deliver behavioral interventions that have been demonstrated as remarkably effective in the social sciences literature on altruism. A patient who participates in the program is assigned a support-sponsor who receives alerts about the patient's adherence, allowing a dialogue of support or problem solving. For the pilot RCT, these support-sponsors will be hired and trained by Keheala. An automated system sends motivational messages and regular prompts for patients to self-verify their treatment. Messages include reminders about the community benefits of adherence and a measure of the patient's adherence performance relative to successful peers. If a patient fails to correctly verify her compliance, the system automatically alerts the support-sponsor, who then intervenes with a supportive dialogue. Clinicians can view individual or aggregate patient histories to leverage limited resources. Combining powerful behavioral interventions with the functionality needed to lessen the burden of disease on everyday life, Keheala uniquely and comprehensively overcomes the barriers to appropriate treatment adherence.

Problem Statement TB treatment adherence rates suffer due to the burdensome six-month duration of treatment. During this period, patients endure severe side effects from drug cocktails, while regular clinical visits often necessitate distant, time-consuming travel and absenteeism from work. However, non-adherence not only threatens the individuals' health--70% of those who aren't treated will die within 10 years --it is also a public health concern: adherence reduces the risk of transmission, usually to nearly zero within less than two weeks, whereas treatment cessation can lead to recurrence and high transmission rates, threatening the well-being of affected communities. Keheala's goal is to increase adherence for the benefit of the infected individual and the community as a whole.

Justification The Keheala solution is based on extensive primary and secondary research. Interviews with relevant and experienced stakeholders ensured that the functionality provided is what actually is needed in order to overcome the social drivers of failed treatment adherence. Additionally, the functionality is designed with principles from the social sciences literature showing the potent impact invoking an individual's sense of responsibility to her community can have on affecting behavior. These principles are well-supported and understood in other contexts, however, exactly how effective these principles can be at invoking treatment adhering behavior in the resource-constrained TB context remains to be tested.

Null Hypotheses Ha1: Patients enrolled in the Keheala program achieve a greater proportion of 'Cured' outcomes by at least 7.5%.

Ho1: Patients enrolled in the Keheala program achieve a greater proportion of 'Cured' outcomes by no more than 7.5%.

Ha2: Patients enrolled in the Keheala program achieve an improvement of at least 7.5% on one of the following outcomes: 'Treatment Completed,' 'Dying while on Treatment,' Out of Control or Loss to Follow Up' and 'Failing'.

Ho2: Patients enrolled in the Keheala program achieve an improvement of no more than 7.5% on one of the following outcomes: 'Treatment Completed,' 'Dying while on Treatment,' Out of Control or Loss to Follow Up' and 'Failing'.

General Objectives The goal of the research is to establish the potential of Keheala's behavioral intervention for positively impacting the process of care and treatment outcomes for a TB patient and healthcare providers.

Additional Qualitative Objectives

* Measure and compare the frequency and duration of treatment interruption
* Measure and compare perception of 'trust' for the healthcare system, as well as the doctor-patient relationship
* Measure and compare the perception of community stigma

Design and Methodology Study site The burden of TB in Kenya is among the highest in the world with a prevalence rate of 558 cases per 100,000 people. Mortality from TB in Kenya is also above the global average at 21 deaths per 100,000.

Symptomatic patients are identified either in health clinics or by Community Health Volunteers (CHVs), laypersons employed to screen for TB in the community. Individuals who show up to the clinic usually do so because they are experiencing a sickness or have been referred to the clinic. In rural communities, regularly scheduled meetings organized by local chiefs or administrative officials are used as opportunities to educate the community about TB and to sometimes distribute questionnaires probing symptoms of TB. Questionnaire respondents who demonstrate signs of symptoms of TB are requested to give a sputum sample, which will be tested at a health clinic and feedback given to the CHV in order to communicate the results back to the individual and link them to a specific clinic if treatment is needed. There are times, however, when finding the individual is not always possible. Additionally, these CHVs will sometimes attend market days or go home to home in order to identify sick individuals in the general population.

Symptoms of TB include coughing for three weeks or longer, chest pain, coughing up blood or sputum (phlegm from deep inside the lungs), weakness or fatigue, weight loss, appetite suppression, fever and chills. Diagnosis is accomplished with sputum smears and sometimes x-rays. Any individuals started on TB medication are entered into a paper log at each health facility. Sub-county TB coordinators compile all of the paper logs every one to four weeks, transferring them to a cloud-based digital form.

Treatment duration is either six months (first-time patients) or eight months (repeat patients). During the first two to three months when daily treatment is required, medications are given for a week at a time or with special permission for longer than a week. For the latter four or five months of treatment patients are required to return to the clinic every two weeks for medication refills. Patients are supposed to visit clinics for medication refills with their treatment supporter - a friend or relative who watches the patient take their medication. However, clinicians do not go to the full-extent necessary to ensure the sponsor has been observing a patient's adherence. Follow-up smears are given after two, five and six months for patients who were initially smear positive. Upon completion of the prescribed treatment regimen and a negative sputum smear, patients are released from treatment and told only to come back if symptoms reappear.

Procedures

The investigators will approach clinics in Nairobi in order of size. Clinics will be included if there is substantial support for the program by the staff and the investigators believe the intervention can be implemented with local support. The investigators will be randomizing subjects into a treatment and control group within each clinic. The following clinics will be approached:

1. Kasarani Health Centre
2. St. Mary's Mission Hospital
3. Riruta Health Centre
4. Kangemi Health Centre
5. Kibera South (MSF Belgium) Dispensary
6. Kayole II Sub-District Hospital
7. Dandora II Health Centre
8. Baraka Medical Centre (St. Stephen)
9. Mukuru MMM Clinic
10. Rhodes Chest Clinic
11. Embakasi Health Centre
12. Ngara Health Centre (City Council of Nairobi)
13. Umoja Health Centre
14. Kibera DO
15. Mathare North Health Centre
16. Kahawa West Health Centre
17. Kamiti Prison Public Hospital (not for inmates)

At each clinic, 50% of all TB patients will be randomly selected to join the treatment group:

* Existing patients will be ordered by date and time admitted, and selected so that every other patient is included in the treatment group (block design).
* New patients will be similarly selected so that every other new patient is included in the treatment group (block design).

The control and treatment groups will thus each be made up of half the patients in the clinics. Overall, the investigators expect the control and treatment group to be comprised of 600 subjects, each. Patients will not be offered a stipend for participation so as not to introduce any unnecessary bias into the study.

Data Management A. Data collection and reduction Clinics will provide paper or digital copies of patient medical records for Keheala staff to consolidate and digitize. Anonymous platform usage data and analytics will be obtained from a dashboard.

Qualitative data will be obtained from a digitally administered survey across the mobile platform and/or through focus group discussions and interviews.

B. Statistical Analysis The simplest possible statistical approach is illustrated in the power calculations. In this approach, the investigators simply compare outcome rates at the end of treatment for subjects in the treatment and control groups. This comparison can be done using a t-test or using an ordinary least squares regression, which can include controls for time trends, patient demographics, and clinic characteristics.

The investigators will also employ a more sophisticated (and slightly more statistically powerful) analysis of hazard rates. The hazard rate is estimated daily as the probability that a patient who is currently adhering continues to adhere. It is estimated using a logistical regression of whether the patient adhered on a given week on whether the patient adhered in all previous weeks and whether the patient is in the treatment group. The regression can also include controls for time period, patient demographics, and clinic characteristics. Note that the investigators have based the power calculations on the simpler regressions of final outcomes on treatment.

C. Data Storage During the study patient names and clinics are kept in an encrypted and password protected 'Master Document'. At the end of the pilot, all personal identifying information will be redacted and patients will be uniquely identified by a randomly generated identification number. No documents or data containing patient identifying information (name and/or address) will be available to outside parties.

Ethical Considerations

The investigators recognize that dealing with human subjects necessitates the highest level of respect for persons. Accordingly, in order to ensure the autonomy of the individual, each patient will receive a full disclosure of the nature of the study, the risks, benefits and alternatives, with an extended opportunity to ask questions. Patients with diminished autonomy (children) will not be coerced to participate. Instead, they will be duly protected through co-consent of the parent and child. No patient will be permitted to participate in the study without having signed an Informed Consent waiver.

The investigators have given forethought to the maximization of benefits and reduction of risks that might occur from the research. The equitable selection and fairness in distribution of participants is only limited by funding; no benefit to which a person is entitled is denied without good reason or when some burden is imposed unduly.

Study limitations As with any study of this nature, focusing on a particular subset of clinics, and excluding some patients limits the generalizability of the results to the population at large (external validity). However, our within-clinic randomization procedure ensures robust internal validity and maximizes statistical power, so that we can maximize the value of this assessment.

Further, the study is limited to a single treatment group, making it impossible to tease apart the impact of Keheala's various elements, evaluate different messages, or different frequency of contact. This decision was made to streamline logistics--these questions are left for a follow-up assessment.

Study Implications A successful pilot would demonstrate the potential of Keheala's low-cost mobile platform to increase compliance and save lives. The investigator's goal is to demonstrate this potential, and also to learn from the implementation in order to maximize the impact of future iterations of the platform.

TB is a particularly ripe use-case for Keheala's platform due to onerous and extended treatment, the limits of existing programs (e.g., the WHO's DOTS program), TB's highly infectious nature, the risk of disease-resistant strains, and its severity. However, Keheala could eventually be applied to address other public health concerns, such as HIV, which shares many of these features. A successful pilot would pave the way for such applications.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with TB by smear microscopy, culture or Gene Xpert.
* Communicate in either Swahili or English.
* Already have access to a mobile phone.

Exclusion Criteria:

- Diagnosed with a drug-resistant strain of TB.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1190 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Unsuccessful Treatment Outcomes | One year
  The proportion of individuals who failed to successfully complete the treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allcott, H. (2011). Social norms and energy conservation. Journal of Public Economics, 95(9), 1082-1095.
- [Background] Andreoni, J., Rao, J. M., & Trachtman, H. (2011). Avoiding the ask: a field experiment on altruism, empathy, and charitable giving (No. w17648). National Bureau of Economic Research.
- [Background] Ayres, I., Raseman, S., & Shih, A. (2013). Evidence from two large field experiments that peer comparison feedback can reduce residential energy usage. Journal of Law, Economics, and Organization, 29(5), 992-1022.
- [Background] Gehlbach, H., Brinkworth, M. E., King, A., Hsu, L., McIntyre, J., & Rogers, T. T. (2015). Creating birds of similar feathers: Leveraging similarity to improve teacher-student relationships and academic achievement.
- [Background] Gollwitzer, P. M. (1999). Implementation intentions: strong effects of simple plans. American psychologist, 54(7), 493.
- [Background] Hallsworth, M., List, J. A., Metcalfe, R. D., & Vlaev, I. (2015). The Making of Homo Honoratus: From Omission to Commission (No. w21210). National Bureau of Economic Research.
- [Background] Hewstone M, Rubin M, Willis H. Intergroup bias. Annu Rev Psychol. 2002;53:575-604. doi: 10.1146/annurev.psych.53.100901.135109. PMID 11752497
- [Background] Karlin B, Zinger JF, Ford R. The effects of feedback on energy conservation: A meta-analysis. Psychol Bull. 2015 Nov;141(6):1205-27. doi: 10.1037/a0039650. Epub 2015 Sep 21. PMID 26390265
- [Background] Knutsson, M., Martinsson, P., & Wollbrant, C. (2013). Do people avoid opportunities to donate?: A natural field experiment on recycling and charitable giving. Journal of Economic Behavior & Organization, 93, 71-77.
- [Background] Kraft-Todd, G., Yoeli, E., Bhanot, S., & Rand, D. (2015). Promoting cooperation in the field. Current Opinion in Behavioral Sciences, 3, 96-101.
- [Background] Malhotra, N., Michelson, M. R., Rogers, T., & Valenzuela, A. A. (2011). Text messages as mobilization tools: The conditional effect of habitual voting and election salience. American Politics Research, 39(4), 664-681.
- [Background] Prestwich A, Perugini M, Hurling R. Can the effects of implementation intentions on exercise be enhanced using text messages? Psychol Health. 2009 Jul;24(6):677-87. doi: 10.1080/08870440802040715. PMID 20205020
- [Background] Rand, D. G., Yoeli, E., & Hoffman, M. (2014). Harnessing reciprocity to promote cooperation and the provisioning of public goods. Policy Insights from the Behavioral and Brain Sciences, 1(1), 263-269.
- [Background] Rege, M., & Telle, K. (2004). The impact of social approval and framing on cooperation in public good situations. Journal of public Economics, 88(7), 1625-1644.
- [Background] Research Center, Pew (2014, February 13). Emerging Nations Embrace Internet, Mobile Technology. Retrieved December 23, 2015, from http://www.pewglobal.org/2014/02/13/emerging-nations-embrace-internet-mobile-technology/
- [Background] Rodgers A, Corbett T, Bramley D, Riddell T, Wills M, Lin RB, Jones M. Do u smoke after txt? Results of a randomised trial of smoking cessation using mobile phone text messaging. Tob Control. 2005 Aug;14(4):255-61. doi: 10.1136/tc.2005.011577. PMID 16046689
- [Background] Rogers, T., Milkman, K., John, L., & Norton, M. I. (2013). Making the best-laid plans better: how plan making increases follow-through. Cambridge, MA: Work. Pap., Harvard Univ.
- [Background] Spranca, M., Minsk, E., & Baron, J. (1991). Omission and commission in judgment and choice. Journal of experimental social psychology, 27(1), 76-105.
- [Background] TB ARC - Centre for Health Solutions. (n.d.). Retrieved 2015, from http://www.chskenya.org/what-we-do/tb-arc/
- [Background] Tiemersma EW, van der Werf MJ, Borgdorff MW, Williams BG, Nagelkerke NJ. Natural history of tuberculosis: duration and fatality of untreated pulmonary tuberculosis in HIV negative patients: a systematic review. PLoS One. 2011 Apr 4;6(4):e17601. doi: 10.1371/journal.pone.0017601. PMID 21483732
- [Background] Tola HH, Tol A, Shojaeizadeh D, Garmaroudi G. Tuberculosis Treatment Non-Adherence and Lost to Follow Up among TB Patients with or without HIV in Developing Countries: A Systematic Review. Iran J Public Health. 2015 Jan;44(1):1-11. PMID 26060770
- [Background] Tuberculosis. (2015, October 1). Retrieved December 12, 2014, from http://www.who.int/mediacentre/factsheets/fs104/en/
- [Background] WHO. (2014). Global Tuberculosis Report 2014. World Health Organization.
- [Background] WHO. (2015). Global Tuberculosis Report 2015. World Health Organization.
- [Background] Yoeli E, Hoffman M, Rand DG, Nowak MA. Powering up with indirect reciprocity in a large-scale field experiment. Proc Natl Acad Sci U S A. 2013 Jun 18;110 Suppl 2(Suppl 2):10424-9. doi: 10.1073/pnas.1301210110. Epub 2013 Jun 10. PMID 23754399
- See also: Keheala - A mobile health platform that uses behavioral interventions to improve healthcare access and treatment outcomes. — https://www.keheala.com/